CLINICAL TRIAL: NCT06729918
Title: The Effect of Virtual Reality-based Learning Tool on Nursing Students' Affective Awareness, Empathy, Self-confidence in Clinical Decision Making and Anxiety Levels
Brief Title: The Effect of Virtual Reality on Affective Awareness, Empathy, Clinical Decision Making in Nursing Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Esra DOĞAN YILMAZ, PhD (Other)
Responsible Party: Sponsor-Investigator, Esra DOĞAN YILMAZ, PhD, Assistant Professor, Kırıkkale University
Organization: Kırıkkale University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: virtual reality-2024
Record Dates: First submitted 2024-12-07; First posted 2024-12-12 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Virtual Reality; Physical Examination of the Thorax and Lungs; Emotional Awareness; Empathy; Self-confidence in Clinical Decision Making and Anxiety
Keywords: virtual reality; physical examination; affective awareness; empathy; self-confidence in clinical decision making and anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: A randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: Data will be entered into the study by someone other than the researchers. Statistical analysis will be performed by someone other than the researchers. Due to the nature of the study, participants will know which group they are in. Therefore, blinding of participants will not be possible. The implementation of the study and collection of data will be performed by the researchers. Therefore, the researchers were not blinded to the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- virtual reality group (Experimental): Thoracic lung physical examination will be studied using a virtual reality-based thoracic and lung physical examination learning tool.
  Interventions: Other: Virtual reality
- simulated patient group (Experimental): Thoracic lung physical examination will be studied using a simulated patient.
  Interventions: Other: simulated patient
- control (traditional education) group (No Intervention): No applicationwas madeto the control group. He/she will practice the thoracic lung physical examination on a classmate who is not in the sample group.

INTERVENTIONS:
Other: Virtual reality — Thoracic lung physical examination will be studied using a virtual reality-based thoracic and lung physical examination learning tool.
  Other Names: Virtual reality based training
  Arms: virtual reality group
Other: simulated patient — Thoracic lung physical examination will be studied using a simulated patient.
  Other Names: simulated patient group
  Arms: simulated patient group

SUMMARY:
This study was planned to be conducted in a randomized controlled experimental design to determine the effect of virtual reality-based learning tool on nursing students' affective awareness, empathy, self-confidence and anxiety levels in clinical decision making. The population of the study will consist of students taking the Health Assessment course at Kırıkkale University, Faculty of Health Sciences, Department of Nursing. The data of the study will be collected by using descriptive characteristics form, "Affective Awareness Scale for Teaching", "Affective and Cognitive Empathy Scale", "Clinical Decision Making Self-Confidence and Anxiety Scale in Nursing". Students will be divided into virtual reality group, simulated patient group and control (traditional education) group using their academic grade point average. The subject of Health Assessment Thorax and Lung assessment will be taught to the control group with traditional education, to the virtual reality group with a virtual reality-based thorax and lung physical examination learning tool, and to the simulated patient group by performing a physical examination of the thorax and lung. Before the application, at the end of the application and at the end of clinical practices, the Affective Awareness Scale for Teaching", 'Affective and Cognitive Empathy Scale', Clinical Decision Making in Nursing Self-Confidence and Anxiety Scale" will be collected. Frequency distributions, descriptive statistics, chi-square, one-way analysis of variance (OneWay ANOVA), Levene's test, "multiple comparison test" (Bonferroni, Tamhane's T2) and repeated measures analysis of variance will be used to evaluate the data. 0.05 will be used as the significance level and it will be stated that there is a significant difference in case of p<0.05 and there is no significant difference in case of p>0.05.

DETAILED DESCRIPTION:
This research will be conducted in a randomized controlled experimental design. This study was planned to determine the effect of virtual reality-based learning tool on nursing students' affective awareness, empathy, self-confidence in clinical decision making and anxiety levels.

Hypothesis 1. Virtual reality-based learning tool affects students' affective awareness Hypothesis 2. Virtual reality-based learning tool affects students' empathy levels.

Hypothesis 3. Virtual reality-based learning tool affects students' self-confidence and anxiety levels in clinical decision making.

The population of the study will consist of 106 student nurses taking the Health Assessment course at Kırıkkale University, Faculty of Health Sciences, Department of Nursing. The sample of the study will consist of students who agree to participate in the study and meet the inclusion criteria.

Randomization in the study; students who meet the sample selection criteria will be randomly divided into 3 groups as virtual reality group, simulated patient group and control (traditional education) group using a computer-based program (www.random.org). Assignment to the virtual reality group, simulated patient group and control (traditional education) groups will be made by an independent researcher to prevent bias and ensure confidentiality.

The data of the study will be collected by using descriptive characteristics form, "Affective Awareness Scale for Teaching", "Affective and Cognitive Empathy Scale", "Self-Confidence and Anxiety Scale for Clinical Decision Making in Nursing".

Descriptive Characteristics Form The "Descriptive Characteristics Form" was developed by the researchers based on the literature.

"Affective Awareness Scale for Teaching" is a scale developed by Yakar and Duman in 2017. The Affective Awareness Scale for Teaching is a 5-point Likert-type scale (1-Not at all suitable for me; 2-Not suitable for me; 3-Suitable for me; 4-Somewhat suitable for me; 5-Completely suitable for me) consisting of five factors: receiving (7 items), reacting (9 items), valuing (8 items), organizing (7 items), and personification (6 items) and a total of 37 items. The Cronbach Alpha reliability coefficient for the overall scale is α=0.896.

"Affective and Cognitive Empathy Scale" is a scale developed by Vachon and Lynam in 2015. The Turkish validity and reliability of the Affective and Cognitive Empathy scale was conducted by Yukay Yüksel et al. in 2020. The Affective and Cognitive Empathy Scale is a scale developed to measure the affective and cognitive levels of participants. This scale allows the researcher to determine the empathy levels of individuals more comprehensively by examining three different empathy dimensions. The Cronbach Alpha reliability coefficient of the scale is α=0.91.

Self-Confidence and Anxiety Scale for Clinical Decision Making in Nursing was developed by Krista A. White in 2014. Turkish validity and reliability was conducted by Bektaş et al. in 2017. The scale evaluates nursing students' anxiety and self-confidence in clinical decision making. The six-point Likert-type scale has a total of 27 questions. Scores are obtained separately for self-confidence and anxiety. As the scores obtained from the self-confidence section and its sub-dimensions increase, the student's self-confidence level increases, and as the scores obtained from the anxiety section and its sub-dimensions decrease, the anxiety level decreases. The lowest score that can be obtained from the self-confidence and anxiety sections is 27 and the highest score is 162. The total Cronbach alpha of the self-confidence section of the scale is 0.97 and the total Cronbach alpha of the anxiety section is 0.96.

Research Implementation The theoretical content of the subject will be explained to all students by the researcher using lecture and question and answer techniques. The students will be administered a descriptive characteristics form, Affective Awareness Scale for Teaching", "Affective and Cognitive Empathy Scale and Self-Confidence and Anxiety Scale for Clinical Decision Making in Nursing (pre-test). Then, students will be randomized into groups according to their academic grade point average.

The virtual reality-based thorax and lung physical examination learning tool was prepared by Aslı Yılmaz and Nurcan Çalışkan. Yılmaz and Çalışkan prepared voice-over content and sound effects to be used in the simulation. After these processes were completed, the algorithm required for the software was created. The researcher planned how the users would move in the simulation, how the menus and controls would work, and how the simulation would respond to the user's actions, and delivered them to the software team. The simulation was developed by the software team using the free and open source "Unity" program to be compatible with the "Oculus" platform.

The simulated patient who will take part in the application was determined. The simulated patient is adult and male. An informative meeting about the process will be held with the simulated patient one week before and on the day of the implementation. Expectations from the simulated patient will be explained at the meeting. Rehearsals will be made regarding the functionality of the application steps and the performance of the simulated patient.

All students in the control group will practice thorax and lung examination on a classmate.

In the health assessment course, three groups will be directed to the laboratories simultaneously. An instructor will be in charge of each group and will ensure coordination. Students in the simulated patient group will work with the simulated patient, students in the virtual reality group will work with virtual reality, and students in the active control group will work on the thorax and lung examination on a classmate who is not in the sample group. While the students are working on the steps of the thorax and lung examination, the instructors will be with them as facilitators. After the practice, the Affective Awareness Scale for Teaching, Affective and Cognitive Empathy Scale, and the Self-Confidence and Anxiety Scale for Clinical Decision Making in Nursing (post-test) will be administered.

During the fall semester of the academic year, students rotate to different clinics (internal and surgical clinics) 2 days a week. At the end of the 15-week fall semester, students will be administered the Affective Awareness Scale for Teaching, Affective and Cognitive Empathy Scale, and the Self-Confidence and Anxiety Scale for Clinical Decision Making in Nursing (follow-up test).

Frequency distributions, descriptive statistics, chi-square, one-way analysis of variance (OneWay ANOVA), Levene's test, "multiple comparison test" (Bonferroni, Tamhane's T2) and repeated measures analysis of variance will be used to evaluate the data. 0.05 will be used as the significance level and it will be stated that there is a significant difference in case of p<0.05 and there is no significant difference in case of p>0.05.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the research
* Not having eye defects that can affect depth perception such as amblyopia (lazy eye), anisometropia (when the refractions of the two eyes are different from each other) and strabismus (strabismus) (The declaration of the person will be taken as basis)
* Having enrolled in the HEM2005 coded "Health Assessment" course for the first time in the Fall Semester of the 2024-2025 Academic Year.

Exclusion Criteria:

* Participation in the research is voluntary
* Graduated from high school, associate degree or undergraduate degree in a health-related field,
* Having taken the HEM2005 coded "Health Assessment" course before were the exclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2024-12-11 (Actual); Primary Completion 2024-12-17 (Actual); Study Completion 2025-01-17 (Actual)

PRIMARY OUTCOMES:
Affective Awareness Level | From the pre-test before the training applications to the post-test after the training applications, approximately one month.
  Scores from sub-dimensions and the scale total are evaluated according to the minimum and maximum scores that can be obtained.
  As the score increases, the level of affective awareness towards teaching also increases.
  Receiving sub-dimension: min: 7, max: 35 Reacting: min: 9, max: 45 Valuing: min: 8, max: 40 Organizing: min: 7, max: 35 Personalizing: min: 6, max: 30 Scale Total Score: min: 37, max: 185
Affective and Cognitive Empathy Level | From the pre-test before the training applications to the post-test after the training applications, approximately one month.
  As the score increases, the level of affective and cognitive empathy also increases.
Clinical Decision Making Self-Confidence and Anxiety Level | As the score increases, the level of affective and cognitive empathy also increases. From the pre-test before the training applications to the post-test after the training applications, approximately one month.
  As the score obtained from the self-confidence section and its sub-dimensions increases, the student's self-confidence level increases, and as the score obtained from the anxiety section and its sub-dimensions decreases, the anxiety level decreases.

CONTACTS AND LOCATIONS:
Overall Officials: Emel GÜLNAR, Assoc. Prof., Principal Investigator — Kırıkkale University; Aslı YILMAZ, MSc, Study Chair — Gazi University graduate student; Esra DOĞAN YILMAZ, Asst. Prof., Study Chair — Kırıkkale University; Kamile KIRCA, Asst. Prof., Study Chair — Kırıkkale University; Şule BIYIK BAYRAM, Assoc. Prof., Study Chair — Black Sea Technical University; Nurcan ÇALIŞKAN, Prof. Dr., Study Chair — Gazi University
Locations (1):
- Kirikkale University, Kırıkkale, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The confidentiality of the data used in the study will be protected.